CLINICAL TRIAL: NCT05982574
Title: Tumor Microenvironment in Lung Adenocarcinoma
Brief Title: Tumor Microenvironment
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. med. Seyer Safi, PD Dr. Seyer Safi, University Hospital Heidelberg
Other Study IDs: S-515/2013 S-270/2001
Record Dates: First submitted 2023-07-30; First posted 2023-08-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer immunotherapy has the great potential to achieve long-term survival in patients with a solid malignancy. However, the beneficial effect of cancer immunotherapy is seen in only a minority of patients. Mounting evidence suggests that immunosuppressive features in the tumor microenvironment prevent an effective antitumor defense. The aim of the investigators is to comprehensively analyze the cytokine profile and the tumor immune infiltrate in the tumor microenvironment and to investigate its prognostic significance in patients with radically resected lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Lung adenocarcinoma
* Tumor stage IB and II
* With or without adjuvant therapy
* Complete surgical resection (R0)
* No distant metastasis at the time of surgery (M0)

Exclusion Criteria:

• Second cancer within 5 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with completely resected lung adenocarcinoma stage IB and II
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of surgery until the date of death from any cause assessed up to 100 months
  Association of tumor microenvironment with overall survival

SECONDARY OUTCOMES:
Recurrence-free survival | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Association of tumor microenvironment with recurrence-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Seyer Safi, MD, Principal Investigator — Technical University of Munich

REFERENCES:
- [Result] Beck C, Ramanujam D, Vaccarello P, Widenmeyer F, Feuerherd M, Cheng CC, Bomhard A, Abikeeva T, Schadler J, Sperhake JP, Graw M, Safi S, Hoffmann H, Staab-Weijnitz CA, Rad R, Protzer U, Frischmuth T, Engelhardt S. Trimannose-coupled antimiR-21 for macrophage-targeted inhalation treatment of acute inflammatory lung damage. Nat Commun. 2023 Jul 28;14(1):4564. doi: 10.1038/s41467-023-40185-1. PMID 37507393
- [Result] Safi S, Messner L, Kliebisch M, Eggert L, Ceylangil C, Lennartz P, Jefferies B, Klein H, Schirren M, Dommasch M, Lobinger D, Multhoff G. Circulating Hsp70 Levels and the Immunophenotype of Peripheral Blood Lymphocytes as Potential Biomarkers for Advanced Lung Cancer and Therapy Failure after Surgery. Biomolecules. 2023 May 22;13(5):874. doi: 10.3390/biom13050874. PMID 37238744
- [Result] Safi S, Yamauchi Y, Hoffmann H, Weichert W, Jost PJ, Winter H, Muley T, Beckhove P. Circulating Interleukin-4 Is Associated with a Systemic T Cell Response against Tumor-Associated Antigens in Treatment-Naive Patients with Resectable Non-Small-Cell Lung Cancer. Cancers (Basel). 2020 Nov 24;12(12):3496. doi: 10.3390/cancers12123496. PMID 33255425